CLINICAL TRIAL: NCT02340104
Title: An Absolute Bioavailability Study of Baricitinib in Healthy Subjects Using the Intravenous Tracer Method
Brief Title: A Study to Measure Baricitinib (LY3009104) Absorption in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14610; I4V-MC-JAGM (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Baricitinib (Experimental): Single oral dose of baricitinib and single intravenous (IV) infusion of [^13C4D3^15N]-baricitinib over 1.5 hours.
  Interventions: Drug: Baricitinib; Drug: [^13C4D3^15N]-baricitinib

INTERVENTIONS:
Drug: Baricitinib — 4 milligrams (mg) administered orally
  Other Names: LY3009104
Drug: [^13C4D3^15N]-baricitinib — 4 micrograms (μg) administered intravenously (IV)
  Other Names: [^13C4D3^15N]-LY3009104

SUMMARY:
The purpose of this study is to compare how much baricitinib (study drug) gets into the blood stream when it is given as a single dose (in tablet form) and as an intravenous infusion (injection given directly into a vein via a small needle). Each participant in the study will make four visits to the investigator site over the course of about 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination
* Male participants: agree to use 2 reliable methods of birth control with female partners of childbearing potential during the study and for at least 3 months following the last dose of study drug
* Female participants: women not of childbearing potential due to surgical sterilization (at least 3 months after surgical hysterectomy, bilateral oophorectomy with or without hysterectomy, or bilateral tubal occlusion/ligation) confirmed by medical history, or menopause. Menopausal women are women with spontaneous amenorrhea for at least 12 months, not induced by a medical condition such as anorexia nervosa and not taking medications during the amenorrhea that induced the amenorrhea (eg, oral contraceptives, hormones, gonadotropin releasing hormone, anti estrogens, selective estrogen receptor modulators, or chemotherapy). Menopausal status should be confirmed by a follicle stimulating hormone (FSH) level greater than 40 international units per liter (IU/L) at screening. Female participants who have been sterilized by tubal ligation will be required to use contraception from the time of screening until 28 days after the last dose of study drug
* Have a body mass index of 18.0 to 32.0 kilogram per meter square (kg/m^2), inclusive, at screening
* Have venous access sufficient to allow for blood sampling and (IV) administration of study drug

Exclusion Criteria:

* Are participants who have previously completed or withdrawn from this study or any other study investigating baricitinib, and have previously received baricitinib
* Have known allergies to baricitinib, related compounds, or any components of the formulation, or history of significant atopy
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a history or presence of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Have a current or recent history (<30 days prior to screening and/or <45 days prior to day before study drug administration) of a clinically significant bacterial, fungal, parasitic, viral (not including rhinopharyngitis), or mycobacterial infection
* Have had symptomatic herpes zoster or herpes simplex infection within 90 days prior to dosing
* Have an absolute neutrophil count (ANC) less than 2 × 109/liter (L) (2000 cells per microliter [cells/μL]) at screening or day before study drug administration. For abnormal values, a single repeat will be allowed
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C infection and/or positive hepatitis C antibody
* Show evidence of hepatitis B infection and/or positive hepatitis B surface antigen
* Are women who are pregnant or lactating
* Have been exposed to a live vaccine within 12 weeks prior to the first dose or expected to need/receive a live vaccine (including herpes zoster vaccination) during the course of the study
* Intend to use over-the-counter or prescription medication and/or herbal supplements within 14 days prior to dosing and during the study (with the exception of occasional paracetamol, which will be permitted at the discretion of the investigator), or intended use of vitamin supplements from study drug administration until discharge from the Clinical Research Unit (CRU)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY, Leeds, Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Baricitinib: Single oral dose of 4 mg baricitinib on Day 1 and approximately the same time a single intravenous (IV) infusion of 4 µg [^13C4D3^15N]-baricitinib over 1.5 hours.
Period: Overall Study
Arm/Group | Baricitinib
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Single oral dose of 4 mg baricitinib on Day 1 and at the same time a single intravenous (IV) infusion of 4 µg [^13C4D3^15N]-baricitinib over 1.5 hours.
Arm/Group | All Participants
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 8

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Baricitinib Following Both the Oral and the IV Dose
Description: AUC[0-∞] is is the area under the concentration verses time curve from zero to infinity, reported as nanograms times hour per milliliter (ng*h/mL).
Time Frame: Predose, 0.5, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 Hours Postdose
Population: All participants who received at least 1 dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Baricitinib Oral Dose: Single oral dose of 4 mg baricitinib
- [^13C4D3^15N]-Baricitinib IV: Single intravenous (IV) infusion of 4 µg[^13C4D3^15N]-baricitinib over 1.5 hours
Arm/Group | Baricitinib Oral Dose | [^13C4D3^15N]-Baricitinib IV
Number analyzed (Participants) | 8 | 8
ng*h/mL | 216 (27) | 0.274 (29)
Statistical Analysis 1: Comparison: Baricitinib Oral Dose vs [^13C4D3^15N]-Baricitinib IV; Test type: Equivalence — Geometric Least Square (LS) Means values were calculated using Log pharmacokinetic (PK) model with treatment, participant, random error as model with treatment as a fixed effect and participant and error as random effects; Ratio of Geometric LS Means = 0.789, 90% CI 2-sided [0.769 to 0.810] — Geometric Least Square (LS) Means values were calculated using Log pharmacokinetic (PK) model with treatment, participant, random error as independent variables, where participant was fitted as a random effect

ADVERSE EVENTS:
Groups:
- Baricitinib: Single oral dose of 4 mg baricitinib on Day 1 and at the same time a single intravenous (IV) infusion of 4 µg [^13C4D3^15N]-baricitinib over 1.5 hours
Arm/Group | Baricitinib
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baricitinib (N=8)
Fatigue (General disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days